CLINICAL TRIAL: NCT05746312
Title: A Digital Music-based Mindfulness Intervention for Elevated Race-based Anxiety in the Black Community: a Replication and Extension
Brief Title: Music-based Mindfulness Intervention for Elevated Race-based Anxiety in the Black Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Grant Jones, Principal Investigator, Harvard University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0256
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: We recruited 8 Black American adults to participate in this multiple baseline study. In a multiple-baseline design, one takes repeated measurements of one's outcomes of interest across time, and subsequently compares these outcomes of interest between an initial baseline control period with no intervention and a subsequent intervention period. This is a within-subjects study design for which participants serve as their own control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple-baseline study (Experimental): All participants in this study received the same protocol. First, we had a baseline control period (no intervention) during which we assessed state anxiety levels every two minutes. Subsequently, we administered the intervention and continued to assess state anxiety at two minute intervals. Participants were randomized to baseline periods that varied in length (10,12,14, or 16 minutes of baseline).
  Interventions: Behavioral: healing attempt

INTERVENTIONS:
Behavioral: healing attempt — The intervention consists of pre-composed and pre-recorded guided meditations, songs, and poems that total 25 minutes in duration. The elements of the intervention were set to background music tracks that were informed by Black diasporic music traditions and anxiety reduction principles from the music therapy literature.

SUMMARY:
This study uses a multiple-baseline design and aims to replicate findings that a digital music-based mindfulness intervention can reduce elevated race-based state anxiety in Black Americans.

ELIGIBILITY:
Inclusion Criteria:

* Familiarity with meditation
* Turns to music for emotional support
* Elevated trait anxiety (>=12 on the State Trait Anxiety Inventory - Trait [STAIT]-5)
* Majority of anxiety comes from racism or discrimination (>=60 on a scale of 0 [not at all] to 100 [entirely] for the following question; "If you are a racial or ethnic minority, how much do you feel that racism and/or discrimination contribute to your elevated anxiety levels?")."

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
State anxiety | Duration of study visit (60-90 minutes)
  Assessed with the State-Trait Anxiety Inventory - 6 [Higher Score = More Anxiety]

CONTACTS AND LOCATIONS:
Overall Officials: Grant Jones, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States